CLINICAL TRIAL: NCT01458730
Title: Immunochemotherapy in Primary Central Nervous System Lymphoma With Rituximab, HD-MTX, HD-Ara C, Cyclophosphamide, Ifosfamide, Vincristine, Vindesine, Temozolomide and DepoCyte Induction Followed by Maintenance Treatment in Elderly Patients With Temozolomide.
Brief Title: Nordic Study in Newly Diagnosed Primary Central Nervous System (CNS) Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Nordic Cancer Union (Other); Roche Pharma AG (Industry); Mundipharma Pte Ltd. (Industry); Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT No 2006-004772-12
Record Dates: First submitted 2011-09-15; First posted 2011-10-25 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Central Nervous System Lymphoma
Keywords: PCNSL; Immunochemotherapy; Intraspinal Depocyt; Maintenance temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Immunochemotherapy — Rituximab, HD-MTX, HD-Ara C, Cyclophosphamide, Iphosphamide, Vincristin, Vindesin, Temozolomide, Depocyte

SUMMARY:
The purpose of the study is to test the efficacy and tolerability of a multiagent chemotherapy treatment regimen without radiotherapy in patients with newly diagnosed lymphoma in the brain.

DETAILED DESCRIPTION:
The objective of the study is

1. To investigate the efficacy and safety of a high-dose methotrexate-based induction polychemotherapy regimen combined with Rituximab and intraspinal DepoCyte followed by temozolomide maintenance treatment in newly diagnosed primary central nervous system lymphoma
2. To assess the long term outcome concerning neurotoxicity

ELIGIBILITY:
Inclusion Criteria:

* Pathologically verified primary central nervous system lymphoma No prior PCNSL treatment.
* Patients treated with steroids alone are eligible
* No signs of lymphoma outside the CNS
* ECOG performance status 0-4
* Age > 17 and < 76 years
* Written informed consent from the patient or guardian

Exclusion Criteria:

* Cardiac failure > 3
* Pregnancy or lactation. Women of childbearing potential are requested to use an effective method of contraception to avoid pregnancy for a period from entry to the study and at least 3 months after the last study medication
* Previous malignancy unless disease free for at least five years
* Active infection.
* Regarding tuberculosis, patients at risk should be tested for latent TB according local practice at each treating centre.
* Positive HIV status
* Organ transplantation
* Serious psychiatric illness
* Prior radiotherapy to the brain
* Concomitant anti-inflammatory medication that cannot be discontinued
* Creatinine clearance < 60 ml/minute calculated by Cockcroft and Gault formula
* Peripheral blood count with granulocytes <1.5 x 109L or platelets < 100 x 109L
* Serum bilirubin >1.5 times or ASAT and alkaline phosphatase >2 times upper limits of normal.
* Known anaphylaxis or IgE-mediated hypersensitivity to murine protein or any component of Rituximab excludes patients from Rituximab treatment, but not from the remaining part of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-05; Primary Completion 2010-10 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Overall survival

SECONDARY OUTCOMES:
response rate | at completion of therapy
neurotoxicity | 1-10 years after completion of therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Elisa Jacobsen Pulczynski, Aarhus, Denmark

REFERENCES:
- [Derived] Pulczynski EJ, Kuittinen O, Erlanson M, Hagberg H, Fossa A, Eriksson M, Nordstrom M, Ostenstad B, Fluge O, Leppa S, Fiirgaard B, Bersvendsen H, Fagerli UM. Successful change of treatment strategy in elderly patients with primary central nervous system lymphoma by de-escalating induction and introducing temozolomide maintenance: results from a phase II study by the Nordic Lymphoma Group. Haematologica. 2015 Apr;100(4):534-40. doi: 10.3324/haematol.2014.108472. Epub 2014 Dec 5. PMID 25480497